CLINICAL TRIAL: NCT03463421
Title: A Prospective Assessment of Adherence and Persistence to Oral Anticoagulation in Ischemic Stroke Patients With Atrial Fibrillation: Incidence, Predictors and the Prognostic Role of the SAMe-TT2R2 Score.
Brief Title: Αdherence and Persistence to Oral Anticoagulation in ΑF Patients With Previous Ischemic Stroke
Acronym: ADHERE-OAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, George Ntaios, MD, MSc (ESO Stroke Medicine), PhD, FESO, Assistant Professor of Internal Medicine, Medical School, University of Thessaly, Larissa University Hospital, University of Thessaly
Other Study IDs: ERISTA 2016
Record Dates: First submitted 2018-02-21; First posted 2018-03-13 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Ischemic Stroke
Keywords: Adherence to oral anticoagulation; Persistence to oral anticoagulation; AF patients; Previous ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aims of this project are to:

1. investigate the adherence and persistence to anticoagulation (and in specific, to VKAs and NOACs) in AF patients with previous ischemic stroke;
2. identify predictors of poor adherence and persistence and
3. assess whether the SAMe-TT2R2 score predicts adherence and persistence to anticoagulation

DETAILED DESCRIPTION:
Patients with ischemic stroke and atrial fibrillation (AF) have a high risk of stroke recurrence, which is the highest among all other pathogenetic subtypes of stroke. This risk is substantially reduced with anticoagulant treatment. For many decades, vitamin-K antagonists (VKA) were the only anticoagulant choice for these patients. However, a number of limitations such as narrow therapeutic window, need for frequent INR measurements and consequent dose adjustments, risk of haemorrhagic complications, food-drug and drug-drug interactions, and others, have undermined the use of anticoagulation by both patients and physicians with apparent influence on the risk of stroke recurrence. During the last decade, four non-vitamin K antagonist oral anticoagulants (NOAC) have been successfully introduced and showed superior safety and efficacy profile than VKAs, more convenient dosing schemes (i.e. no need for adjustments) and minimum interactions with food and drugs. These advantages of NOACs vs. VKAs may have obvious implications to patient adherence to treatment and, consequently, to the efficacy of secondary stroke prevention. Nevertheless, there are only very scarce data available yet that the adherence and persistence to NOACs is higher than the adherence and persistence to VKAs in the specific population of patients with ischemic stroke and atrial fibrillation.

Recently, the SAMe-TT2R2 score has been introduced as a means to identify those AF patients who have inadequate quality of anticoagulation with VKAs expressed as Time within Therapeutic Range (TTR)5. In specific, VKA-anticoagulated AF patients with a SAMe-TT2R2 score of 0-2 are expected to have a TTR >65%, whereas patients with a score of >2 are expected to have lower TTR levels. In this context, one could hypothesize that increased SAMe-TT2R2 score may be associated with inadequate adherence and persistence to VKAs. Other parameters associated with inadequate adherence and persistence in the general AF population include education, employment, social status, and cognitive function. However, this is not well investigated in the specific population of patients with previous stroke where other conditions such as age and functional neurological status may also play an important role in adherence and persistence.

ELIGIBILITY:
Inclusion Criteria:

* Previous ischemic stroke
* Atrial fibrillation
* Age >18 years
* Informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The dataset will be derived mainly from two high quality, prospective stroke registries: the Larissa Stroke Outcome Registry (LASTRO)(Larissa University Hospital, Greece) and the Helsinki Stroke Registry (Helsinki University Hospital, Finland)
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Adherence to medication | Up to 5 years
  The Adherence to Refills and Medications Scale (ARMS) will be used to assess adherence to medication. The ARMS consists of 12 items, each one representing a 4-point question. It was also designed to include two distinct subscales, and this was supported in the overall factor analysis. The 8-item medication taking subscale assesses a patient's ability to correctly self-administer the prescribed regimen. The 4-item prescription refill subscale assesses a patient's ability to refill medications on schedule. Conceptually, these represent different types of problems in medication use In the publication that introduced the ARMS score (Kripalani et al. Value Health. 2009 Jan-Feb;12(1):118-23), on the eight-item taking medications subscale, scores ranged from 8 to 29 (mean = 10.33, SD = 2.66), and in the four-item refilling medications subscale, scores from 4 to 14 were reported (mean = 5.99, SD = 1.98). Lower scores indicate better adherence.

SECONDARY OUTCOMES:
Proportion of patients still on the initial anticoagulant at the time of follow-up assessment | Up to 5 years
  Persistence to oral anticoagulation

CONTACTS AND LOCATIONS:
Overall Officials: George Ntaios, MD, PhD, Principal Investigator — Medical School, University of Thessaly, Larissa University Hospital
Locations (2):
- Department of Neurology, Helsinki University Hospital, Helsinki, FinlandHelsinki University Hospital, Helsinki, Finland
- Medical School, University of Thessaly, Larissa University Hospital, Larissa, Greece

IPD SHARING:
Plan to Share IPD: Undecided